CLINICAL TRIAL: NCT02466841
Title: Prospective Comparison of Techniques for Cubital Tunnel Release
Status: Withdrawn | Type: Observational
Why Stopped: Could not get any patients to sign up
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, John Fowler, MD, University of Pittsburgh
Other Study IDs: PRO15040063
Record Dates: First submitted 2015-06-03; First posted 2015-06-09 (Estimated); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Cubital Tunnel Syndrome
MeSH Terms: conditions — Cubital Tunnel Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients undergoing cubital tunnel release surgery: Patients undergoing cubital tunnel release surgery will be enrolled. All enrolled subjects will be followed regardless of the technique used by surgeon.
  Interventions: Procedure: Cubital tunnel release

INTERVENTIONS:
Procedure: Cubital tunnel release — Patients undergoing cubital tunnel release for ulnar nerve compression at elbow

SUMMARY:
Compression of the ulnar nerve at the elbow (cubital tunnel syndrome) is the second most common compressive neuropathy of the upper extremity (carpal tunnel is the most common). Patients who fail conservative treatment (activity modification, splinting, medications) are offered cubital tunnel release. There are multiple techniques to decompress the ulnar nerve at the elbow, but the ideal release has not been determined. These techniques vary from simple decompression of the nerve (in-situ release, endoscopic release), to decompressing the nerve and moving it anteriorly to take tension off the nerve (subcutaneous transposition, sub-fascial transposition, sub muscular transposition), and removing part of the medial epicondyle (medial epicondylectomy). Each procedure has purported benefits and also potential complications. Simple in-situ release has the benefit of shorter operative times and less surgical dissection, however, the nerve may subluxate post-operatively and cause persistent pain. Procedures to move the nerve (subcutaneous transposition, sub-fascial transposition, sub muscular transposition) prevent subluxation and take tension off the nerve, however, they require more dissection, larger incisions, and also partially devascularize the nerve. Medial epicondylectomy prevents subluxation and decompresses the nerve, but some patients may have a prolonged recovery and persistent pain from removing part of the bone.

The purpose of this study is to prospective evaluate patients undergoing cubital tunnel release according to the standard practice and preference of their surgeon. The investigators plan to compare the different techniques at standard post-operative intervals.

DETAILED DESCRIPTION:
Objective:

The purpose of this study is to compare different techniques for cubital tunnel release.

Specific Aims:

1. Determine if there are differences in patient-directed outcomes scores between different techniques used for cubital tunnel release.
2. Determine if there are differences in post-operative pain scores between different techniques used for cubital tunnel release.
3. Determine if there are differences in objective measurements such as range of motion and grip strength scores between different techniques used for cubital tunnel release.
4. Determine if there are differences in complications between different techniques used for cubital tunnel release.

Background:

Compression of the ulnar nerve at the elbow (cubital tunnel syndrome) is the second most common compressive neuropathy of the upper extremity (carpal tunnel is the most common). Patients who fail conservative treatment (activity modification, splinting, medications) are offered cubital tunnel release. There are multiple techniques to decompress the ulnar nerve at the elbow, but the ideal release has not been determined. These techniques vary from simple decompression of the nerve (in-situ release, endoscopic release), to decompressing the nerve and moving it anteriorly to take tension off the nerve (subcutaneous transposition, sub-fascial transposition, sub muscular transposition), and removing part of the medial epicondyle (medial epicondylectomy). Each procedure has purported benefits and also potential complications. Simple in-situ release has the benefit of shorter operative times and less surgical dissection, however, the nerve may subluxate post-operatively and cause persistent pain. Procedures to move the nerve (subcutaneous transposition, sub-fascial transposition, sub muscular transposition) prevent subluxation and take tension off the nerve, however, they require more dissection, larger incisions, and also partially devascularize the nerve. Medial epicondylectomy prevents subluxation and decompresses the nerve, but some patients may have a prolonged recovery and persistent pain from removing part of the bone.

Significance:

The results of this study may provide a high level of evidence to determine if specific techniques for cubital tunnel decompression result in improved patient outcomes and/or fewer complications.

ELIGIBILITY:
Inclusion Criteria:

* patients indicated to surgery by attending surgeon

Exclusion Criteria:

* previous cubital tunnel release on ipsilateral side
* unable/unwilling to provide consent
* pregnant women
* prisoners
* < 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing cubital tunnel release
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-08; Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Patient rated ulnar nerve evaluation (PRUNE) score | 1 year
  The PRUNE is a validated patient rated outcome measurement to assess pain, symptoms and functional disability in patients with ulnar nerve compression at the elbow.

SECONDARY OUTCOMES:
Elbow Range of Motion | 1 year
  The elbow range of motion will be measured in degrees.
Visual Analog Scale (VAS) for Pain | 1 year
  The VAS for pain is a patient-reported single-item scale with scores ranging 0 (no pain) to 10 (worst pain).
2 Point Discrimination Test | 1 year
  The test will measure, in millimeters, the ability of a patient to determine discern the difference between two points when 2 separate instruments are touched to the skin.
Hand Dynamometer to measure Grip Strength | 1 year
  The Hand Dynamometer is a simple hand-held device when squeezed, will report grip strength in kgs.
Number of subjects with post-surgical complications | 1 year
  The presence or absence of post-surgical complications will be recorded for each subject.

REFERENCES:
- [Background] Palmer BA, Hughes TB. Cubital tunnel syndrome. J Hand Surg Am. 2010 Jan;35(1):153-63. doi: 10.1016/j.jhsa.2009.11.004. PMID 20117320
- [Background] Osei DA, Padegimas EM, Calfee RP, Gelberman RH. Outcomes following modified oblique medial epicondylectomy for treatment of cubital tunnel syndrome. J Hand Surg Am. 2013 Feb;38(2):336-43. doi: 10.1016/j.jhsa.2012.11.006. Epub 2013 Jan 3. PMID 23291082
- [Background] MacDermid JC, Grewal R. Development and validation of the patient-rated ulnar nerve evaluation. BMC Musculoskelet Disord. 2013 Apr 26;14:146. doi: 10.1186/1471-2474-14-146. PMID 23617407